CLINICAL TRIAL: NCT05870176
Title: ActivityChoice: A Clinic-delivered Implementation Program to Increase Physical Activity and Decrease Cardiovascular Disease Risk Amongst Cancer Survivors
Brief Title: ActivityChoice: Implementing Clinic-Based Physical Activity Program Choices for Cancer Survivors
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jamie Faro, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000522; 1K01HL163254 (NIH)
Record Dates: First submitted 2023-05-01; First posted 2023-05-23 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Cardiovascular Diseases; Physical Inactivity
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Stepped-wedge sequential crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Referral (Active Comparator): Provider education/training on referral process Patient education material on physical activity benefits Paper referral to LIVESTRONG at the YMCA Fitbit Activity Monitor
  Interventions: Behavioral: Standard Referral
- Enhanced Referral (Experimental): Provider education/training on referral process Patient education material on physical activity benefits Patient decision aid on physical activity program choices Electronic referral to program of patient's choice Fitbit Activity Monitor
  Interventions: Behavioral: Enhanced Referral

INTERVENTIONS:
Behavioral: Enhanced Referral — The enhanced referral uses an electronic referral and patient decision aid to provide choices to 3 different physical activity programs.
  Arms: Enhanced Referral
Behavioral: Standard Referral — The standard referral period will serve as the "usual care" comparator. Patients will receive a paper referral and Fitbit monitor.
  Arms: Standard Referral

SUMMARY:
Cardiovascular disease, the number one leading cause of death in the United States, is highly prevalent in cancer survivors. Physical activity can reduce risk, and referrals to programs addressing survivors' choices are highly recommended from providers in cancer survivorship, though rarely implemented. The study team proposes to develop ActivityChoice, a clinic-based implementation program, using patient narrative decision aids to support choices to a group in-person, group virtual, or self-monitored digital health physical activity program.

ELIGIBILITY:
AIM 1 Inclusion Criteria for Aim 1a

1. Prior cancer diagnosis
2. 18 years of age and older
3. Speaks English

Exclusion Criteria for Aim 1a

1. No prior cancer diagnosis
2. Under 18 years of age
3. Prisoners
4. Does not speak English

AIM1B Survivor Inclusion Criteria for Aim 1b

1. Prior cancer diagnosis
2. 18 years of age and older
3. Speaks English

Survivor Exclusion Criteria for 1b

1. No prior cancer diagnosis
2. Under 18 years of age
3. Does not speak English
4. Prisoners
5. Participated in Aim 1a

Clinic Staff Inclusion Criteria for Aim 1b

1. Provide cancer care for patients at one of the four UMass cancer clinics,
2. Involved in survivorship care planning visits
3. Speaks English
4. 18 years of age and older

Clinic Staff Exclusion Criteria for 1b

1. Is not employed at one of the four UMass cancer clinics
2. Is not involved in survivorship care planning visits
3. Does not speak English
4. Prisoners
5. Under 18 years of age

Pregnant Women Pregnant women may be included in this study as an incidental population.

AIM 2 Clinic Staff Inclusion Criteria for Aim 2

1. Provide cancer care for patients at one of the four UMass cancer clinics
2. Involved in survivorship care visits
3. Speaks English
4. 18 years of age and older

Clinic Staff Exclusion Criteria for Aim 2

1. Is not employed at one of the four UMass cancer clinics
2. Is not involved in survivorship care visits
3. Does not speak English
4. Prisoners
5. Under 18 years of age

Survivor Inclusion Criteria for Aim 2

1. Cancer Patient at one of the four UMass cancer clinics
2. Has a survivorship care planning visit
3. Able to perform physical activity
4. Completes Physical Activity Readiness Questionnaire (PAR-Q) physical activity readiness questionnaire or has medical clearance to participate
5. Has a smartphone
6. Speaks English
7. 18 years of age and older

Survivor Exclusion Criteria for Aim 2:

1. Not a cancer patient at one of the four UMass cancer clinics
2. Does not have a survivorship care planning visit
3. Unable to perform physical activity or no medical clearance to participate
4. Does not speak English
5. Under 18 years of age
6. Does not have a smartphone
7. Prisoners
8. Is pregnant

AIM 3 Clinic Staff Inclusion Criteria for Aim 3

1. Are enrolled in ActivityChoice
2. ≥ 18 years of age
3. Provide written informed consent

Patient Inclusion Criteria for Aim 3

1. Are enrolled in ActivityChoice
2. Had a clinic visit with one of the enrolled clinic staff during the study period
3. ≥ 18 years of age
4. Speaks English
5. Provide written informed consent

Patient Exclusion Criteria for Aim 3

1. Not enrolled in ActivityChoice
2. Was not seen in the clinic by an enrolled clinic staff during the study period

UMass Cancer Clinic Administration Inclusion Criteria for Aim 3

1. Are ≥ 18 years of age
2. Are in positions of cancer center leadership
3. Provide written informed consent

UMass Cancer Clinic Administration Exclusion Criteria for Aim 3

1. Unable or unwilling to provide written informed consent
2. Not in positions of leadership within the UMass Medical Cancer Clinic Administration
3. <18 years of age.

External site stakeholders Inclusion Criteria for Aim 3

1. Are ≥18 years of age
2. Are in positions of cancer center leadership
3. Provide written informed consent.

External site stakeholders Exclusion Criteria for Aim 3

1. Unable or unwilling to provide written informed consent
2. Not in positions of leadership overseeing cancer survivorship
3. <18 years of age.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients referred as obtained by the electronic referral system and electronic health record | Baseline
  The number of patients referred/The number of eligible patients

SECONDARY OUTCOMES:
Proportion of eligible clinicians enrolling in the the study | Baseline
  Number of enrolled clinicians/Number of eligible clinicians
Clinic/Clinician fidelity of delivering patient decision aids | Baseline
  Clinic delivery of patient decision aids as reported by patients
Patient Engagement | Examined at baseline, 3-, and 6-months
  Program enrollment (number referred/number enrolled);
Patient Retention | 3- and 6-months
  Percent of enrolled patients completing follow-up surveys at 3- and 6-months
Patient narrative decision aid acceptability and effectiveness (Enhanced Referral only) | Baseline following referrals
  Acceptability of decision aid using the Ottawa Decision Aid Centre 10-item acceptability of decision aids (Minimum score=0, Maximum score=100; Higher score indicates higher decisional conflict and uncertainty
Patient Autonomous Regulation | Baseline, 3- and 6-months
  Behavioral Regulation for Exercise Questionnaire-2 (Minimum=0, Maximum=76; Higher scores indicates greater regulation/motivation)
Patient Objective Physical Activity | Baseline, 3- and 6-months
  Change from baseline to 3- and 6-months in steps, light, moderate and vigorous physical activity measured via Fitbits.
Patient Self-Report Physical Activity | Baseline, 3- and 6-months
  Change from baseline to 3- and 6-months in light, moderate and vigorous physical activity survey-measured (Godin leisure time questionnaire) physical activity. The questionnaire is a 4-item self-administered questionnaire with the first three questions seeking information on the number of times one engages in mild, moderate and strenuous leisure-time physical activity bouts of at least 15 min duration in a typical week. Scores can range from 0 to 98, with the higher score meaning a greater level of activity for that week.
Patient Health-related Quality of Life | Baseline, 3- and 6-months
  Functional Assessment of Cancer Therapy-General (FACT-G): Physical, social, emotional and functional well-being (Minimum=0, Maximum=127; Higher score means a higher quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Faro, PhD, Principal Investigator — UMass Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No